CLINICAL TRIAL: NCT03261180
Title: Perioperative Nutritional Optimization in Head and Neck Cancer Patients
Brief Title: Nestle Impact Advanced Recovery in Improving Surgery Recovery in Patients With Head and Neck Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniel Clayburgh, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00015929; NCI-2017-01480 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00015929 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Nestle Impact AR) (Experimental): Patients receive Nestle Impact AR for 5 days before and after surgery in addition to regular diet.
  Interventions: Other: Laboratory Biomarker Analysis; Dietary Supplement: Nutritional Intervention
- Group II (regular diet) (Active Comparator): Patients receive regular diet.
  Interventions: Other: Best Practice; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Best Practice — Receive regular diet
  Other Names: standard of care; standard therapy
  Arms: Group II (regular diet)
Other: Laboratory Biomarker Analysis — Correlative studies
Dietary Supplement: Nutritional Intervention — Receive Nestle Impact AR
  Arms: Group I (Nestle Impact AR)

SUMMARY:
This randomized clinical trial studies how well Nestle Impact Advanced Recovery works in improving surgery recovery in patients with head and neck cancer. Adding a nutritional supplement, such as Nestle Impact Advanced Recovery to a regular diet before and after head and neck cancer surgery may help to decrease the number of wound complications after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the effect of perioperative use of Nestle Impact Advanced Recovery (AR) on the rate of post-operative wound complications within 30 days after major head and neck surgery.

SECONDARY OBJECTIVES:

I. Assess whether sarcopenia is an independent risk factor for the development of post-operative wound complications.

II. Assess whether Nestle IMPACT AR decreases the rate of other post-operative complications such as pneumonia, urinary tract infection, deep vein thrombosis, and clostridium difficile colitis within 30 days of surgery, as well as length of hospital stay.

TERTIARY OBJECTIVES:

I. Assess changes in muscle metabolic gene expression at the time of surgery associated with sarcopenia and IMAPCT treatment.

OUTLINE: Patients are randomized into 1 of 2 groups.

GROUP I: Patients receive Nestle Impact AR for 5 days before and after surgery in addition to regular diet.

GROUP I: Patients receive regular diet.

After completion of study, patients are followed up for 30 days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Members of all races and ethnic groups will be included
* Patients must be diagnosed with cancer of the head and neck and must be surgical candidates
* Patients must be indicated for major head and neck surgery, defined as surgeries with an anticipated post-surgical hospital stay of 4 or more days; examples of major surgeries include, but are not limited to, total laryngectomy, large oral cavity, oropharyngeal, salivary gland, or soft tissue resections requiring free flap or major regional flap (e.g. pectoralis major flap), and large skull base procedures requiring extensive skull base reconstruction
* Patients must have cross-sectional body imaging (positron emission tomography [PET]-computed tomography [CT] or equivalent) performed within 4 weeks of study enrollment and available for review
* Patient must be willing to receive Nestle IMPACT Advance Recovery for five days prior to planned surgery as well as for 5 days after surgery
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with known distant metastases or other malignancies
* Patients unable to tolerate oral intake by mouth or per enteral feeding tube
* Patients with galactosemia
* Patients who have received any investigational medication within 6 weeks of enrollment, or who are scheduled to receive an investigational drug during the course of the study
* Patients currently taking IMPACT or other immunonutrition products (arginine-containing supplements) will be excluded; other forms of nutritional supplementation, such as caloric supplementation, tube feeding, or other dietary supplements are allowed on study
* Patients currently taking anabolic steroids will be excluded; patients taking corticosteroids are allowed on study
* Psychiatric illness/social situations that would limit compliance with study requirements
* Excluded patients will be allowed to participate in the trial on an observational basis only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-08-10 (Estimated); Study Completion 2021-08-09 (Estimated)

PRIMARY OUTCOMES:
Rate of post-operative wound complications | Within 30 days after major head and neck surgery
  A patient is found to have a post-operative complication is one of the following is observed: wound infection, seroma, wound dehiscence, fistula formation, free tissue flap loss. A 2-sided 95% confidence interval will also be calculated for each arm, using exact methods, and chi square testing will be performed to compare the incidence of wound complications within 30 days after surgery between control and experimental groups. A multivariate analysis of the primary endpoint will be performed with logistic regression to include study treatment, presence of sarcopenia, prior radiation therapy, a

SECONDARY OUTCOMES:
Rate of other post-operative complications | Within 30 days after surgery
  Will assess whether Nestle IMPACT Advanced Recovery (AR) decreases the rate of other post-operative complications within 30 days after surgery such as pneumonia, urinary tract infection, deep vein thrombosis, and clostridium difficile colitis as well as length of hospital stay. Will be analyzed using chi square testing. The analysis of the length of the stay (LOS) for patients in each arm will be analyzed using the Kaplan Meier method for estimation of summary statistics including the 25th, 50th (median), and 75th percentiles and associated 95% confidence intervals. Patients that die prior to
Sarcopenia | Within 30 days after major head and neck surgery
  Will assess whether sarcopenia is an independent risk factor for the development of 30-day post-operative wound complications. Will be analyzed using chi square testing.

OTHER OUTCOMES:
Sarcopenia-related gene expression | Up to 30 days post-surgery
  Will asses messenger ribonucleic acid expression level of the sarcopenia-related genes MAFbx, MuRF1, Foxo1, Redd1, Sesn1, SELP, IL-6, BNIP3, and CTSL1, within skeletal muscle, and circulating levels of sarcopenia-associated exomes. Will be analyzed using chi square testing.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clayburgh, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States